CLINICAL TRIAL: NCT01618110
Title: Transcranial Magnetic Stimulation of the Pre-Frontal Cortex in the Treatment of Attention Deficit/Hyperactivity Disorders: A Randomized, Controlled, Double Blind Study.
Brief Title: Transcranial Magnetic Stimulation in Treatment of Attention Deficit/Hyperactivity Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH-12-0012
Record Dates: First submitted 2012-06-10; First posted 2012-06-13 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: ADHD; Attention Deficit/Hyperactivity Disorder; TMS; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Magnetic Stimulation; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Active Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation (Magstim, Rapid)
- Sham group (Sham Comparator): Sham TMS coil (same noise, minimal magnetic field)
  Interventions: Other: Placebo Treatment

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (Magstim, Rapid) — Superficial rTMS, directed at right PFC, power of 100% of MT, 10Hz for 4 seconds, intervals of 30 seconds, 42 trains.
  Other Names: Magstim, Rapid; Transcranial Magnetic Stimulation
  Arms: Treatment Group
Other: Placebo Treatment — Sham coil (minimal magnetic field, same noise and feeling)
  Other Names: Placebo; Sham
  Arms: Sham group

SUMMARY:
* ADHD is one of the most common psychiatric disorders.
* While most of the attention is directed towards youth, 60% continue to suffer symptoms into adult life.
* Current treatment is effective, but 30% suffer side effects that lowers QOL, and 20% are non-responders.
* Known mechanism of pathophysiology includes hypoactive dopaminergic system, especially at right PFC.
* It is this study hypothesis that by stimulating the right PFC by TMS, it will be possible to alleviate ADHD symptoms.
* A 10 sessions of treatment will by applied on a randomly allocated group of patients, diagnosed with ADHD, in a 2:1 ratio: The first group will receive an actual TMS treatment, and the second group will receive a sham treatment.
* Improvement of objective and subjective ADHD scale will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Established diagnosis of ADHD
* No C/I for TMS
* Has signed an informed consent form

Exclusion Criteria:

* Major Psychiatric disorders (Psychotic or Affective)
* Active use of drugs (4 weeks prior to participation)
* Neurologic disorder such as Epilepsy.
* No use of stimulants during the previous 7 days

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Bloch, MD, Principal Investigator — Shalvata MHC
Locations (1):
- Shalvata MHC, Hod HaSharon, Israel